CLINICAL TRIAL: NCT05800210
Title: Alpha/Beta T Cell and CD19+ B Cell Depletion in Allogeneic Stem Cell Transplantation in Patients With Malignant Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government); Ocala Royal Dames for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-PED-004
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndromes; Chronic Myeloid Leukemia; Lymphoma, Non-Hodgkin; Lymphoma, Hodgkin
Keywords: hematologic malignancy; GVHD; stem cell transplantation; graft manipulation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Allogeneic stem cell transplant with ⍺/β CD3+ T-cell and CD19+ B-cell depleted graft (Experimental)
  Interventions: Device: Miltenyi CliniMACS Prodigy ® system

INTERVENTIONS:
Device: Miltenyi CliniMACS Prodigy ® system — Subjects will receive an allogeneic stem cell transplant that has been depleted of ⍺/β CD3+ T-cells and CD19+ B-cells using the Miltenyi CliniMACS Prodigy® system.

SUMMARY:
This study will assess the safety, efficacy, and feasibility of ⍺/β CD3+ T-cell and CD19+ B-cell depletion in allogeneic stem cell transplantation in patients with acute lymphocytic leukemia (ALL), acute myeloid leukemia (AML), juvenile myelomonocytic leukemia (JMML), high risk myelodysplastic syndrome (MDS), chronic myeloid leukemia (CML) and lymphoma. Subjects will receive an allogeneic stem cell transplant that has been depleted of ⍺/β CD3+ T-cells and CD19+ B-cells using the Miltenyi CliniMACS Prodigy® system.

ELIGIBILITY:
Inclusion Criteria:

A. Children, Adolescents, Young adults (ages 6 months to ≤39 years) with the following diseases may be eligible:

i. ALL

1. ALL high risk including one or more of the following: (t(9;22) or 11q23 chromosomal abnormality, primary induction failure (≤15% blasts at time of registration), mixed phenotype acute leukemia (MPAL), persistent MRD (≥0.01% by flow or persistent abnormal karyotype detected by cytogenetics) or hypodiploidy (≤44 chromosomes)) in first remission
2. ALL in second remission and beyond

ii. AML

1. History of AML induction/reinduction Failure (≤15% blasts at time of registration)
2. AML in CR1 with poor cytogenetics (i.e., 12p, 5a, -7, FLT3 mutation/duplication, t(9;11) and others)
3. AML with persistent minimal residual disease (MRD) in CR1(≥0.01% on flow or persistent abnormal karyotype detected by cytogenetics)
4. AML CR2 or beyond
5. AML in refractory relapse but ≤15% bone marrow leukemia blasts
6. Therapy-related AML

iii. Juvenile MyeloMonocytic Leukemia (JMML)

1. JMML in CR1 without CBL mutation
2. JMML with recurrence of disease with or without CBL mutation
3. JMML CR2 or beyond

iv. Chronic Myeloid Leukemia (CML)

1. CML in CR with regard to blast crisis

v. High Risk Myelodysplastic syndrome (MDS)

vi. Lymphoma: Hodgkin (HL) or Non-Hodgkin (NHL)

1. HL or NHL with a history of induction failure
2. HL or NHL in PR1 or PR2
3. HL or NHL in CR2 or subsequent remission

B. Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included).

C. HLA-matched (5-6/6) sibling donor, matched (8-10/10) unrelated donor available for stem cell donation, haplo-identical related donor (at least one full haplotype must be matched).

D. Karnofsky or Lansky score ≥60% at the time of enrollment. Karnofsky scores must be used for patients >16 years of age and Lansky scores for patients ≤16 years of age.

E. Adequate organ function (within 4 weeks of initiation of preparative regimen), defined as:

i. Pulmonary: FEV1, FVC, and corrected DLCO must all be ≥ 60% of predicted by pulmonary function tests (PFTs). For children who are unable to perform for PFTs due to age, the criteria are: no evidence of dyspnea at rest and no need for supplemental oxygen.

ii. Renal: Creatinine clearance or radioisotope GFR ≥60 mL/min/1.73 m2 or a serum creatinine based on age/gender

iii. Cardiac: Shortening fraction of ≥ 27% by echocardiogram) or ejection fraction of ≥ 50% by echocardiogram or radionuclide scan (MUGA).

iv. Hepatic: SGOT (AST) or SGPT (ALT) < 5 x upper limit of normal (ULN) for age. Conjugated bilirubin < 2.5 mg/dL, unless attributable to Gilbert's Syndrome.

F. Written informed consent obtained from the subject or guardian and the subject agrees to comply with all the study-related procedures.

G. Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 8 weeks after the last dose of study drug to minimize the risk of pregnancy.

H. Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 8 weeks following the last dose of study drug.

Exclusion Criteria:

A. Patients with documented uncontrolled infection

B. Patients who have received allogeneic hematopoietic stem cell transplantation within 6 months, unless being done as a boost.

C. Patients with active ≥Grade 2 aGVHD.

D. Demonstrated lack of compliance with medical care.

E. Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 8 weeks after the last dose of study drug.

F. Females who are known to be pregnant or breastfeeding.

G. History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.

H. Prisoners or subjects who are incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 6 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Acute graft versus host disease (aGVHD) incidence | 100 days
  Compare the incidence of grade II to IV aGVHD following allogeneic stem cell trasplantation utilizing α/β CD3+ T-cell and CD19+ B-cell depletion compared to historical controls by day +100

SECONDARY OUTCOMES:
Event-free survival | 2 years
  Evaluate the event-free survival, which is defined as being alive and without evidence of disease relapse
Overall survival | 2 years
  Evaluate the overall survival
Probability of hematopoietic engraftment | 100 days
  Determine the probability of hematopoietic engraftment, as measured by the presence of donor chimerism >95% by day 100
Cytomegalovirus (CMV) viremia incidence | 1 year
  Determine the incidence of CMV viremia. Viremia is defined as >1000copies/mL present on at least 2 weekly tests or requiring therapy.
Epstein-Barr virus (EBV) viremia incidence | 1 year
  Determine the incidence of EBV viremia. Viremia is defined as >1000copies/mL present on at least 2 weekly tests or requiring therapy.
Adenovirus viremia incidence | 1 year
  Determine the incidence of adenovirus viremia. Viremia is defined as >1000copies/mL present on at least 2 weekly tests or requiring therapy.
Post-transplant lymphoproliferative disorder (PTLD) incidence | 1 year
  Determine the incidence of PTLD

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Milner, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States